CLINICAL TRIAL: NCT03953092
Title: A Randomized, Double-blind, Placebo-controlled, Sequential Single and Multiple Ascending Doses (SAD/MAD) Study Following Oral Administration in Healthy Subjects to Evaluate the Safety, Tolerability, and Pharmacokinetics of YG1699
Brief Title: A Randomized, Double-blind, Placebo-controlled, Sequential Single and Multiple Ascending Doses of YG1699
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Youngene Therapeutics Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: YG1699 -01
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Diabete Mellitus
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Single Ascending Dose and Multiple Ascending Dose
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- SAD Cohort 1 (Experimental): 5 mg YG1699 or Placebo
  Interventions: Drug: YG1699; Drug: Placebos
- SAD Cohort 2 (Experimental): 10 mg YG1699 or placebo
  Interventions: Drug: YG1699; Drug: Placebos
- SAD Cohort 3 (Experimental): 25 mg YG1699 or placebo
  Interventions: Drug: YG1699; Drug: Placebos
- SAD Cohort 4 (Experimental): 50 mg YG1699 or placebo
  Interventions: Drug: YG1699; Drug: Placebos
- SAD Cohort 5 (Experimental): 100 mg YG1699 or placebo
  Interventions: Drug: YG1699; Drug: Placebos
- MAD Cohort 1 (Experimental): 5 mg YG1699 or placebo
  Interventions: Drug: YG1699; Drug: Placebos
- MAD Cohort 2 (Experimental): 20 mg YG1699 or placebo
  Interventions: Drug: YG1699; Drug: Placebos
- MAD Cohort 3 (Experimental): 50 mg YG1699 or placebo
  Interventions: Drug: YG1699; Drug: Placebos

INTERVENTIONS:
Drug: YG1699 — YG1699 at Multiple Doses
Drug: Placebos — Placebos

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose-escalation study to evaluate the safety, tolerability, and pharmacokinetics (PK) of YG1699 following single and multiple ascending oral dose administration.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, dose-escalation study to evaluate the safety, tolerability, and pharmacokinetics (PK) of YG1699 following single and multiple ascending oral dose administration.

The study consists of 2 parts: Part 1, SAD dose-escalation; Part 2, MAD dose-escalation.

ELIGIBILITY:
Inclusion Criteria:

1. Are capable of giving informed consent and complying with study procedures;
2. Are between the ages of 18 and 55 years, inclusive;
3. Female subjects have a negative urine pregnancy test result at screening and Day -1, and meet one of the following criteria:

   1. Using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives) [e.g., hormonal contraceptives (oral, patch, injectable or vaginal ring), implantable device (implantable rod or intrauterine device), or a double barrier (e.g., diaphragm, cervical cap, oral, patch or vaginal hormonal contraceptive, condom, spermicide, or sponge)]
   2. Surgically sterile for at least 3 months prior to screening by one of the following means:

      * Bilateral tubal ligation
      * Bilateral salpingectomy (with or without oophorectomy)
      * Surgical hysterectomy
      * Bilateral oophorectomy (with or without hysterectomy)
   3. Postmenopausal, defined as the following:

      * Last menstrual period greater than 12 months prior to screening
      * Postmenopausal status confirmed by serum FSH and estradiol levels at screening;
4. Considered healthy by the Investigator, based on subject's reported medical history, full physical examination, clinical laboratory tests, 12-lead ECG, and vital signs;
5. Normal renal function with estimated glomerular filtration rate (eGFR) of 60 ml/min/1.73m2 or greater and as deemed by the Investigator;
6. Non-smoker and no more than 2 tobacco-containing including nicotine replacement products in last 6 months;
7. Body mass index (BMI) of 18.0 to 30.0 kg/m2 inclusive and body weight not less than 50 kg;
8. Willing and able to adhere to study restrictions and to be confined at the clinical research center.
9. Male subjects with female partners of child bearing potential must agree to use condoms for the duration of the study and until 12 weeks after dosing with the study drug and must refrain from donating sperm for this same period.

Exclusion Criteria:

1. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity as determined by the Investigator;
2. Known or suspected malignancy;
3. History of pancreatitis or gall stones;
4. History of unexplained syncope, symptomatic hypotension or hypoglycemia;
5. Family history of long QTc syndrome;
6. History of chronic diarrhea, malabsorption, unexplained weight loss, food allergies or intolerance;
7. Poor venous access;
8. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody;
9. Donated or lost >500ml of blood in the previous 3 months;
10. Taken an investigational drug or participated in a clinical trial within 3 months (or 5 half-lives), whichever is longer;
11. Taken any prescription medications within 14 days or 5 half-lives (whichever is longer) of the first dose of study drug;
12. Hospital admission or major surgery within 6 months prior to screening;
13. A history of prescription drug abuse, or illicit drug use within 9 months prior to screening;
14. A history of alcohol abuse according to medical history within 9 months prior to screening;
15. A positive screen for alcohol, drugs of abuse at screening or Day -1;
16. An unwillingness or inability to comply with food and beverage restrictions during study participation;
17. Use of over-the-counter (OTC) medication within 7 days, and herbal (including St John's Wort, herbal teas, garlic extracts) within 7 days prior to dosing (Note: Use of acetaminophen at < 2 g/day is permitted until 24 hours prior to dosing);
18. Any condition or finding that in the Investigators opinion would put the subject or study conduct at risk if the subject were to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Adverse events will be evaluated | 76 Days
  Safety and Tolerability of YG1699

SECONDARY OUTCOMES:
Area Under the Curve [AUC] | 76 Days
  area under the plasma drug concentration time curve from time 0 to T (AUC)
maximum plasma concentration (Cmax) | 76 days
  maximum plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Yalin Li, MD, Study Director — Youngene Therapeutics Inc., Ltd.
Locations (1):
- Frontage Labs, Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No